CLINICAL TRIAL: NCT00407498
Title: An Open Label Multicentric Phase 1 Study of Selective Cyclin Dependent Kinase Inhibitor P276-00 in Patients With Advanced Refractory Neoplasms
Brief Title: Open Label Phase I Study of P276-00 in Patients With Advanced Refractory Neoplasms
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Piramal Enterprises Limited (Industry)
Responsible Party: Dr Himanshu Parikh, Nicholas Piramal India Limited
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P276-00/01/04
Record Dates: First submitted 2006-12-04; First posted 2006-12-05 (Estimated); Last update posted 2009-01-01 (Estimated); Status verified 2008-12

CONDITIONS: Neoplasm
Keywords: P 276-00; Advanced Refractory Neoplasm; Maximum Tolerated Dose; Dose Limiting Toxicity; Pharmacokinetics
MeSH Terms: conditions — Neoplasms | interventions — P276-00

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: P276-00 — Starting dose of 9 mg/m2/day from day 1to 5 and day 8 to 12 in 21 day cycle.Protocol wa amended to dose the subjects for day 1 to5 in 21 day cycle after 34.4 mg/m2/day cohort.Maximum dose administered was 259 mg/m2/day

SUMMARY:
P276-00 is specific Cdk4-D1 and Cdk1-B inhibitor. P276-00 exhibited significant tumour reduction in animal models with less adverse effects.Based on the results from various in-vitro studies, P276-00 could be a potential candidate as a new mechanism based drug for the treatment of cancer.This Phase I study will determine the Maximum Tolerated Dose,Dose Limiting Toxicity and efficacy of P 276-00 in patients with advanced Refractory neoplasms.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically and/ or cytologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective.
2. Patients of either sex, of all races and ethnic groups, and > 18 years of age
3. ECOG (Eastern Cooperative Oncology Group) performance status < 2
4. Patients with life expectancy of at least 4 months.
5. Patients must have normal organ and marrow function as defined below:

   * absolute neutrophil count ≥ 1,500/mL
   * platelets ≥ 100,000/mL
   * total bilirubin within normal institutional limits
   * AST/ALT ≤ 2.5 X institutional upper limit of normal (ULN)
   * creatinine within 1.5 times the upper normal institutional limits
6. The effects of P276-00 on the developing human foetus are unknown. For this reason women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, during the duration of study participation and for at least 4 weeks after withdrawal from the study.
7. Concomitant medications for diabetes, hypertension, pain relief and any other co-existing conditions, except cancer, are permitted when the patient is on study medication. There should be no change in the dosage of these medications in the 2 weeks prior to day 1 of cycle 1, with the exception of dosages for pain relief medication. Changes in the dose of anti-emetics and diuretics may be made provided they will not interfere with probable adverse effects of investigational product.
8. Ability to understand and the willingness to sign a written informed consent document.
9. Patients must have measurable disease.

Exclusion Criteria:

1. Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study (date of consent); or patients who have not recovered from adverse events (except grade 1 toxicities) due to agents administered more than 4 weeks earlier.
2. Patients having received any other investigational agents within 4 weeks prior to the date of consent and patients who have not recovered completely from the side effects of the earlier investigational agent.
3. Patients with known brain metastases should be excluded from this clinical trial.
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to P276-00.
5. Patients having history of myocardial infarction or uncontrolled cardiac dysfunction during the previous 6 months.
6. Patients having diarrhoea requiring anti-diarrhoeal therapy.
7. Patients with uncontrolled and unstable intercurrent illness.
8. Women who are pregnant or nursing. P276-00 may have the potential for teratogenic or abortifacient effects. Since there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with P276-00, breastfeeding should be discontinued if the mother is to be treated with P276-00.
9. Patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy. Therefore, HIV-positive patients are excluded from the study.
10. Patients requiring the use of concomitant medications that prolong the QT/QTc interval and /or are known to cause Torsades de Pointes (TdP)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-05; Primary Completion 2008-03 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose and dose limiting toxicity of selective Cdk inhibitor P276-00 in patients with advanced refractory neoplasms. | DLT to be seen for cycle 1.Adverse events as and when they occur during the trial duration and till their resolution after exit from study

SECONDARY OUTCOMES:
To determine the toxic effects, pharmacokinetics and clinical response of this regimen. | Pharmacokinetics on day 1 and 5 of cycle 1, clinical response after every 2 cycles, toxic effects of the drug as and when they occur to be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Hal Hirte, MD, FRCP, Principal Investigator — Juravinsky Cancer Centre; Tara Baetz, MD, FRCP, Principal Investigator — Kingston Health Sciences Centre; Raghunadharao D, MD, DM, Principal Investigator — Nizam's Institute of Medicai Sciences
Locations (3):
- Canada (2):
  - Juravinsky Cancer Centre, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
- Nizam's Institute of Medicai Sciences, Hyderabaad, Andhrapradesh, India

REFERENCES:
- [Result] Hirte H.W, Raghunatharao D, Baetz S, Hotte J, Rajappa S, Iaccobucci A, Sharma S, Parikh H, Kulkarni S, Patil S, Padigaru M, Gaston S. A Phase I study of the selective cyclin dependant kinase inhibitor P276-00 in Patients with advanced refractory neoplasms. AACR 2007 Abstract number #802
- [Derived] Malumbres M, Barbacid M. Cell cycle, CDKs and cancer: a changing paradigm. Nat Rev Cancer. 2009 Mar;9(3):153-66. doi: 10.1038/nrc2602. PMID 19238148